CLINICAL TRIAL: NCT02942030
Title: Differences in Attentional Profile of Children Diagnosed With ADHD Versus Children Diagnosed With Other Mental Conditions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 000816-com2
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADHD: Children diagnosed with ADHD after a complete psychiatric evaluation.
  Interventions: Other: Computerized assesment battery
- Non-ADHD: Children diagnosed with other mental conditions after a complete psychiatric evaluation.
  Interventions: Other: Computerized assesment battery

INTERVENTIONS:
Other: Computerized assesment battery — All participants will do a computerized assessment battery to identify specific attentional profile

SUMMARY:
Attentional symptoms characterize both ADHD and other mental conditions in children.

The diagnosis is based on clinical psychiatric evaluation.

With the expanding knowledge regarding the neurobiological basis in ADHD the investigators have learned that attention is not a general property of the whole brain, but involves several coordinated networks. This knowledge promoted the scientific community to the stage in which scientists can recognize different types of attention domains.

in the current study, the investigators use computerized battery to separate between the different attention abilities and provide specific attentional profile. in this study the investigators aim to characterize different attentional profiles in children who are diagnosed with ADHD versus children who diagnosed with other mental condition (which are common differential diagnoses of ADHD)

DETAILED DESCRIPTION:
Attentional symptoms characterize both ADHD and other mental conditions in children.

The diagnosis of ADHD is based on clinical psychiatric evaluation in different clinical situations the differential diagnosis is not straight forward and the clinician considers a common co-morbid conditions and common differential diagnoses.

With the expanding knowledge regarding the neurobiological basis in ADHD the scientific community have learned that attention is not a general property of the whole brain, but involves several coordinated networks. This knowledge promoted us to the stage in which scientists can recognize different types of attention domains. this knowledge raises the question - can the clinician use this knowledge to make the correct diagnosis based on specific attentional profile?

In the current study, the investigators use computerized battery in order to separate between the different attention abilities and provide specific attentional profile. in this study the investigators aim to characterize different attentional profiles in children who are diagnosed with ADHD versus children who diagnosed with other mental condition (which are common differential diagnoses of ADHD)

ELIGIBILITY:
Inclusion Criteria:

* age 8-12
* normal intelligence quotient (IQ)
* suspected ADHD

Exclusion Criteria:

* Autism Spectrum Disorder
* blindness
* deafness
* abnormal intelligence quotient (IQ) (below 70)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 8-12 y/o children reffered to a psychiatric clinic for evaluation
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
diagnosis - after psychiatric evaluation | november 2017
attentional computerized profile | november 2017

SECONDARY OUTCOMES:
correlations - clinical diagnosis and attentional profile | november 2017

CONTACTS AND LOCATIONS:
Overall Officials: shlomit tsafrir, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Mishmar Ha'Am Clinic, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No